CLINICAL TRIAL: NCT06253091
Title: Comparison of the Application of Robot-assisted Laparoscopic Transperitoneal and Transperitoneal Pathways in Radical Cystectomy
Brief Title: Comparison of the Application of Robot-assisted Laparoscopic Pathways in Radical Cystectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-SR-017
Record Dates: First submitted 2024-02-03; First posted 2024-02-12 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Bladder Cancer
Keywords: radical cystectomy
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- robit-assist transperitoneal laparoscopic radical cystectomy (No Intervention): robit-assist radical cystectomy was performed transperitoneal
- robit-assist extraperitoneal laparoscopic radical cystectomy (Experimental): robit-assist radical cystectomy was performed extraperitoneal
  Interventions: Procedure: robit-assist extraperitoneal laparoscopic radical cystectomy

INTERVENTIONS:
Procedure: robit-assist extraperitoneal laparoscopic radical cystectomy — robit-assist laparoscopic radical cystectomy was performed extraperitoneal
  Arms: robit-assist extraperitoneal laparoscopic radical cystectomy

SUMMARY:
Traditional radical cystectomy (RC) is performed transabdominal. However, it often has high postoperative complications. There have been studies on extraperitoneal approach to reduce postoperative complications. Investigators divided participants underwent robot-assisted radical cystectomy into two groups (1:1) . One group of participants transabdominal, the other group extraperitoneal. The incidence of complications and PFS/OS at 3, and 5 years were compared.

DETAILED DESCRIPTION:
Bladder cancer is highly prevalent worldwide and approximately 75% of these are non-muscle invasive bladder cancer (NMIBC). For high-risk NMIBC and MIBC, radical cystectomy (RC) is also the best treatment option.

The traditional transperitoneal laparoscopic radical cystectomy prolapse of abdominal organs into the pelvic cavity can lead to angulation of the intestinal tract, causing obstruction. Some studies have demonstrated that the extraperitoneal route can effectively reduce these complications Currently, robot-assisted surgery technology is widely utilized in urology. Studies have demonstrated that robot-assisted total extraperitoneal cystectomy and urinary diversion are less likely to disrupt abdominal organs, particularly the intestines. Identifying and locating membrane structures and layers with anatomical significance is crucial for navigating the correct anatomic space during the operation. The using of 3D laparoscopy or a robot-assisted extraperitoneal radical cystectomy aligns more closely with the 3D membrane anatomic concept. Furthermore, for younger patients,robot-assisted extraperitoneal radical cystectomy is more favorable for preserving reproductive function. For elderly patients, it is considered more safer.

Consequently, we aim to investigate whether robot-assisted extraperitoneal radical cystectomy is more advantageous for patients with MIBC or high-risk NMIBC.

ELIGIBILITY:
Inclusion Criteria:

1. Researchers evaluated patients with muscle invasive bladder cancer or high-risk non-muscular invasive bladder cancer who needed radical cystectomy.
2. Willing to accept the operation and meet the surgical index: a) Absolute count of neutrophils≥1.5x109/L; b) Platelets≥100×109/L; c) Hemoglobin≥90g/L; d) International standardized ratio or activationPartial thrombin time≤1.5 Upper limit of normal value (ULN); e) calculated creatinine clearance rate≥1 ml/s; f) Total serum bilirubin≤1.5×ULN; g) AST, ALT and alkaline phosphatase≤2.5×ULN; h) Cardiopulmonary function indicates that it can tolerate major abdominal surgery;
3. None of the pastHistory of abdominal surgery;
4. 18 to 75 years old;
5. ECOG physical state 0 or 1;
6. voluntarily participate in this experiment, be able to provide a written version of the informed consent, and be able to understand and agree to comply with the requirements of this study and the evaluation schedule;

Exclusion Criteria:

1. Patients who refuse to receive radical cystectomy
2. Researchers evaluate patients who are unable to tolerate radical cystectomy;
3. There is a abdominal history of surgery;
4. Have had a large-scale operation or major trauma within 28 days before joining the group;
5. Have been vaccinated with live vaccine within 28 days before joining the group;
6. Severe chronic or active infection that requires systemic anti-bacterial, antifungal or antiviral treatment within 14 days before joining the group;
7. Participating in the rest of the clinical research.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Complication rate | through study completion, an average of 1 month, 3 month and 1 year
  Complication rate after surgery

SECONDARY OUTCOMES:
OS | 5 years after surgery
  Overall Survival
PFS | 5 years after surgery
  progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Lv qiang, PhD, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The first affiliated hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lobo N, Afferi L, Moschini M, Mostafid H, Porten S, Psutka SP, Gupta S, Smith AB, Williams SB, Lotan Y. Epidemiology, Screening, and Prevention of Bladder Cancer. Eur Urol Oncol. 2022 Dec;5(6):628-639. doi: 10.1016/j.euo.2022.10.003. Epub 2022 Nov 1. PMID 36333236
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Knowles MA, Hurst CD. Molecular biology of bladder cancer: new insights into pathogenesis and clinical diversity. Nat Rev Cancer. 2015 Jan;15(1):25-41. doi: 10.1038/nrc3817. PMID 25533674
- [Background] Witjes JA, Bruins HM, Cathomas R, Comperat EM, Cowan NC, Gakis G, Hernandez V, Linares Espinos E, Lorch A, Neuzillet Y, Rouanne M, Thalmann GN, Veskimae E, Ribal MJ, van der Heijden AG. European Association of Urology Guidelines on Muscle-invasive and Metastatic Bladder Cancer: Summary of the 2020 Guidelines. Eur Urol. 2021 Jan;79(1):82-104. doi: 10.1016/j.eururo.2020.03.055. Epub 2020 Apr 29. PMID 32360052
- [Background] Haeuser L, Marchese M, Noldus J, Kibel AS, Carvalho F, Preston MA, Cooper Z, Trinh QD, Mossanen M. Association between Operative Time and Short-Term Radical Cystectomy Complications. Urol Int. 2023;107(3):273-279. doi: 10.1159/000522141. Epub 2022 Mar 18. PMID 35306500
- [Background] Parra RO, Andrus CH, Jones JP, Boullier JA. Laparoscopic cystectomy: initial report on a new treatment for the retained bladder. J Urol. 1992 Oct;148(4):1140-4. doi: 10.1016/s0022-5347(17)36843-x. PMID 1404624
- [Background] Cao Q, Li P, Yang X, Qian J, Wang Z, Lu Q, Gu M. Laparoscopic radical cystectomy with pelvic re-peritonealization: the technique and initial clinical outcomes. BMC Urol. 2018 Dec 12;18(1):113. doi: 10.1186/s12894-018-0424-6. PMID 30541538
- [Background] Kulkarni JN, Gulla RI, Tongaonkar HB, Kashyapi BD, Rajyaguru KB. Radical cystoprostatectomy: an extraperitoneal retrograde approach. J Urol. 1999 Feb;161(2):545-8. doi: 10.1016/s0022-5347(01)61946-3. PMID 9915445
- [Background] Zhu YP, Ye DW, Yao XD, Zhang SL, Dai B, Shen YJ, Wang CF. Defining good candidates for extraperitoneal cystectomy: results from random peritoneum biopsies of 136 cases. Urology. 2013 Apr;81(4):820-4. doi: 10.1016/j.urology.2012.11.057. Epub 2013 Feb 20. PMID 23434097
- [Background] Park DS, Gong IH, Choi DK, Hwang JH, Kang MH, Oh JJ. A feasibility study of peritoneum preservation in radical cystectomy with extraperitonealization of orthotopic neobladder for invasive high-grade bladder cancer: a preliminary analysis. Int Urol Nephrol. 2014 Jun;46(6):1107-13. doi: 10.1007/s11255-013-0632-7. Epub 2013 Dec 20. PMID 24356919
- [Background] De Nunzio C, Cicione A, Leonardo F, Rondoni M, Franco G, Cantiani A, Tubaro A, Leonardo C. Extraperitoneal radical cystectomy and ureterocutaneostomy in octogenarians. Int Urol Nephrol. 2011 Sep;43(3):663-7. doi: 10.1007/s11255-010-9876-7. Epub 2010 Nov 26. PMID 21110093
- [Background] Jentzmik F, Schostak M, Stephan C, Baumunk D, Lingnau A, Weikert S, Lein M, Miller K, Schrader M. Extraperitoneal radical cystectomy with extraperitonealization of the ileal neobladder: a comparison to the transperitoneal technique. World J Urol. 2010 Aug;28(4):457-63. doi: 10.1007/s00345-009-0476-z. Epub 2009 Sep 24. PMID 19777243
- [Background] Feng L, Song J, Wu M, Tian Y, Zhang D. Extraperitoneal versus transperitoneal laparoscopic radical cystectomy for selected elderly bladder cancer patients: a single center experience. Int Braz J Urol. 2016 Jul-Aug;42(4):655-62. doi: 10.1590/S1677-5538.IBJU.2015.0608. PMID 27564274
- [Background] Refaai K, Sharafeldin MA, Elabbady A, Sameh W, Thurairaja R, Nair R, Dasgupta P, Khan MS, Mohamed E. Perioperative Outcomes of Open Retrograde Extraperitoneal Versus Intracorporeal Robot-assisted Radical Cystoprostatectomy in Men: A Dual-center Comparative Study. Clin Genitourin Cancer. 2020 Jun;18(3):e315-e323. doi: 10.1016/j.clgc.2019.12.006. Epub 2019 Dec 14. PMID 31911120
- [Background] Kulkarni JN, Agarwal H. Transperitoneal vs. extraperitoneal radical cystectomy for bladder cancer: A retrospective study. Int Braz J Urol. 2018 Mar-Apr;44(2):296-303. doi: 10.1590/S1677-5538.IBJU.2017.0441. PMID 29219280
- [Background] Zhao J, Zeng S, Zhang Z, Zhou T, Yang B, Song R, Sun Y, Xu C. Laparoscopic Radical Cystectomy Versus Extraperitoneal Radical Cystectomy: Is the Extraperitoneal Technique Rewarding? Clin Genitourin Cancer. 2015 Aug;13(4):e271-e277. doi: 10.1016/j.clgc.2015.01.006. Epub 2015 Jan 21. PMID 25743207
- [Background] Zhu G, Zhang Z, Zhao K, Yin X, Zhang Y, Wang Z, Li C, Sui Y, Li X, Yang H, Xing N, Wang K. Laparoscopic radical cystectomy with pelvic lymph node dissection and ileal orthotopic neobladder by a total extraperitoneal approach: Our initial technique and short-term outcomes. Investig Clin Urol. 2022 Sep;63(5):523-530. doi: 10.4111/icu.20220156. PMID 36067997
- [Background] Soleimani M, Moradkhani E, Masoumi N, Gholivandan J. Extra-Peritoneal versus Trans-Peritoneal Open Radical Cystectomy - Comparison of Two Techniques in Early Post-Operative Complications. Urol J. 2021 Nov 7;18(5):519-524. doi: 10.22037/uj.v16i7.6147. PMID 32827149
- [Background] Yang H, Zhang Z, Zhao K, Zhang Y, Yin X, Zhu G, Lin C, Liu C, Wang Z, Sui Y, Li X, Li C, Wang K. Extraperitoneal Laparoscopic Radical Cystectomy With Preservation of Fertility for the Treatment of Ewing Sarcoma: The First Report of a Reliable Surgical Method. Urology. 2022 Jan;159:241-246. doi: 10.1016/j.urology.2021.09.024. Epub 2021 Oct 13. PMID 34653432
- [Background] Malinaric R, Mantica G, Balzarini F, Terrone C, Maffezzini M. Extraperitoneal cystectomy with ureterocutaneostomy derivation in fragile patients - should it be performed more often? Arch Ital Urol Androl. 2022 Jun 29;94(2):144-149. doi: 10.4081/aiua.2022.2.144. PMID 35775336
- [Background] Li Z, Zhang Z, Ma H, Yao K, Qin Z, Han H, Ye Y, Li Y, Dong P, Jiang L, Tian L, Liu Z, Zhou F. Extraperitonealization of ileal conduit reduces parastomal hernia after cystectomy and ileal conduit diversion. Urol Oncol. 2022 Apr;40(4):162.e17-162.e23. doi: 10.1016/j.urolonc.2021.11.022. Epub 2021 Dec 15. PMID 34920945
- [Background] Kulkarni JN, Rizvi SJ, Acharya UP, Kumar KS, Tiwari P. Gynecologic-tract sparing extra peritoneal retrograde radical cystectomy with neobladder. Int Braz J Urol. 2008 Mar-Apr;34(2):180-7; discussion 187-90. doi: 10.1590/s1677-55382008000200008. PMID 18462516